CLINICAL TRIAL: NCT06903663
Title: A Multi-Centric, Retrospective, Real-World Study on First-Line Therapy With Atezolizumab Plus Bevacizumab for Advanced or Unresectable Hepatocellular Carcinoma in Romanian Population
Brief Title: The Epidemiology of Patients Treated With ATZ+BEV in Real Life Setting
Acronym: MANIFEST-HCC
Status: Not yet recruiting | Type: Observational
Sponsor: Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor (Other)
Collaborators: MDX Research (Network)
Responsible Party: Principal Investigator, Adrian Radu Vidra, Lead Investigator Adrian Radu Vidra, MD, Senior Specialist in Medical Oncology, Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor
Other Study IDs: MANIFEST-HCC-RO
Record Dates: First submitted 2025-02-12; First posted 2025-04-01 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Descriptive epidemiology of patients treated with ATZ plus BEV; Pathological features of HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult women and men (≥ 18 years of age) with proven initial diagnosis of HCC: Patients with HCC following treatment with ATZ plus BEV identified from the patient registry in the hospital with treatment charts between April 1, 2022- December 31, 2024 (index date).

SUMMARY:
Hepatocellular carcinoma (HCC) is the sixth most prevalent cancer and the third most frequent cause of cancer-related death globally.

This retrospective, multicentric study will be coordinated by Dr. Adrian Radu Vidra (Lead Investigator) from Regional Institute of Gastroenterology and Hepatology "Prof. Dr. Octavian Fodor" Cluj-Napoca (Coordinating Site) to further investigate the clinical and demographic profile of patients receiving first-line treatment with atezolizumab and bevacizumab in the real-world setting of clinical practice from Romania.

Participants already taking the combination therapy as part of their regular medical care for HCC will be followed during 3 years.

DETAILED DESCRIPTION:
The available information suggests that the ATZ plus BEV is safe and effective as first-line systemic therapy for patients with unresected HCC and advanced HCC. The overall efficacy and safety of the combination has been well established in the literature and from the various clinical studies. This combination has since replaced tyrosine kinase inhibitors as the standard for many patients. The combination significantly increases OS (median 19.2 months vs. 13.4 months with sorafenib) and objective response rates (30% vs. 11%), offering better disease control.

The defined primary study outcome is describing the epidemiology of patients treated with ATZ+BEV in real-life setting.

History of the disease, including etiology of liver disease, BCLC stage, MVI, EHS, Child-Pugh Score, ALBI grade, MELD, Betablocker medication, Prior treatment, Resection, Local ablation, TACE/SIRT, BMI, ALT, AST, TBL, Albumin, INR, AFP will be collected and presented.

Data on baseline characteristics, radiological response, treatment patterns and adverse events will be summarized using descriptive statistics. Continuous variables will be presented shown as median and full range, and categorical variables will be reported as frequencies and percentages.

Median duration of therapy was defined as the time from the first administration until the last administration of the drugs. Patients who still received atezolizumab with or without concomitant bevacizumab at data cut-off will be censored.

Patients with at least one staging imaging assessment will be evaluated for radiological response.

Data from patients, who died without radiologically confirmed tumor progression, will be censored at the date of the last radiological assessment or death.

PFS is defined as the time from the date of the first therapy administration until radiological disease progression or death, whatever occurred first. Patients still alive and without radiologically confirmed progression at the date of the last contact or data cut-off will be censored.

OS will be defined as the time from the start of the treatment with atezolizumab and bevacizumab until the date of death.

Survival curves will be calculated with the Kaplan-Meier method and compared by means of the log-rank test.

Safety assessment will consist of monitoring the incidence of all adverse events observed following the treatment with ATZ plus BEV, graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5. Safety events will be stratified by type of events, grades, seriousness and will be collected at time points defined in the study flowchart.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women and men (≥ 18 years of age) with proven initial diagnosis of HCC with evidence of loco-regional recurrent or advanced disease not amenable to resection.
2. At least one cycle of therapy with ATZ plus BEV.
3. Eligible individuals will be required to have Baseline (pre-index) EGD available
4. No prior systemic therapy for HCC.
5. Evaluable disease as defined per modified Response Evaluation Criteria in Solid Tumours (mRECIST) V1.1 criterion (At least 1 evaluable CT result over the entire available index and post-index period, excluding the baseline).
6. Patients identified from the patient registry in the hospital with treatment charts between April 1, 2022- December 31, 2024 (index date).
7. Eligible individuals will be required to have data available prior to the index date (pre-index period; baseline characteristics).

Exclusion Criteria:

1. A diagnosis of any other primary cancer prior to the index date
2. ATZ plus BEV treatment as part of a clinical trial
3. ATZ or BEV given off-label
4. Patients with incomplete medical records
5. Patients receiving other investigational drugs
6. History of hepatic encephalopathy
7. Patients with brain metastasis
8. HBV and HBC co-infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with a diagnosis of advanced or unresectable HCC undergoing combined therapy with atezolizumab and bevacizumab.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Description of the epidemiology of patients treated with ATZ+BEV | 36 months
  The defined primary study outcome is describing the epidemiology of patients treated with ATZ+BEV in real life setting.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) according to viral and non-viral etiology in the selected cohort | 36 months
  PFS is defined as the time from the date of the first therapy administration until radiological disease progression or death, whatever occurred first. Patients still alive and without radiologically confirmed progression at the date of the last contact or data cut-off will be censored.
Overall Survival (OS) for patients treated with the combination therapy | 36 months
  OS will be defined as the elapsed time from onset of the treatment to death from any cause. For surviving patients, follow-up will be censored at the date of last contact (or last date known to be alive). Follow-up for OS will be performed at 12, 24, 30, 36 months (3.0 years).
Disease Control Rate (DCR) | 36 months
  DCR will be calculated per modified Response Evaluation Criteria in Solid Tumors (mRECIST) V1.1 criterion, as the proportion of patients with best overall response to protocol therapy of complete response (CR), partial response (PR) or stable disease (SD) that is maintained for at least 12 weeks.
Objective Response Rate (ORR) | 36 months
  ORR will be defined as the proportion of the patients with a confirmed CR or PR, as per mRECIST V1.1 criterion.
Duration of Response (DOR) | 36 months
  DOR will be defined as the elapsed time from documented tumor response to documented disease progression or death from any cause.
Overall safety of the combined therapy | 36 months
  Safety assessment will consist of monitoring the incidence of all adverse events observed following the treatment with ATZ plus BEV, graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5. Safety events will be stratified by type of events, grades, seriousness and will be collected at time points defined in the study flowchart.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Radu Vidra, Principal Investigator — Regional Institute of Gastroenterology and Hepatology "Prof. Dr. Octavian Fodor" Cluj-Napoca
Locations (4):
- Romania (4):
  - Fundeni Clinical Institute, Bucharest, Bucharest
  - Regional Institute of Gastroenterology and Hepatology "Prof. Dr. Octavian Fodor", Cluj-Napoca, Cluj
  - Regional Institute of Oncology, Iași, Iaşi
  - Oncohelp, Timișoara, Timiș County

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kulkarni AV, Tevethia H, Kumar K, Premkumar M, Muttaiah MD, Hiraoka A, Hatanaka T, Tada T, Kumada T, Kakizaki S, Vogel A, Finn RS, Rao PN, Pillai A, Reddy DN, Singal AG. Effectiveness and safety of atezolizumab-bevacizumab in patients with unresectable hepatocellular carcinoma: a systematic review and meta-analysis. EClinicalMedicine. 2023 Aug 30;63:102179. doi: 10.1016/j.eclinm.2023.102179. eCollection 2023 Sep. PMID 37680945
- [Background] Storandt MH, Zemla TJ, Patell K, Naleid N, Gile JJ, Tran NH, Chakrabarti S, Jin Z, Borad M, Mahipal A. Atezolizumab plus bevacizumab as first-line systemic therapy for hepatocellular carcinoma: a multi-institutional cohort study. Oncologist. 2024 Nov 4;29(11):986-996. doi: 10.1093/oncolo/oyae142. PMID 38979643
- [Background] Bialecki ES, Di Bisceglie AM. Diagnosis of hepatocellular carcinoma. HPB (Oxford). 2005;7(1):26-34. doi: 10.1080/13651820410024049. PMID 18333158
- [Background] Pinero F, da Fonseca LG. Trial eligibility in advanced hepatocellular carcinoma: Does it support clinical practice in underrepresented subgroups? World J Gastroenterol. 2021 Jun 28;27(24):3429-3439. doi: 10.3748/wjg.v27.i24.3429. PMID 34239261
- [Background] Singal AG, Ozgurdal K, Fan X, Vassilev Z, Pan X, Multani JK, Chen CC, Zhou Z, He J, Pisa F. Real-World Systemic Treatment Patterns after Atezolizumab and Bevacizumab in Patients with Hepatocellular Carcinoma in the United States. Cancers (Basel). 2023 Nov 22;15(23):5532. doi: 10.3390/cancers15235532. PMID 38067235
- [Background] Cheng AL, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Lim HY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Ma N, Nicholas A, Wang Y, Li L, Zhu AX, Finn RS. Updated efficacy and safety data from IMbrave150: Atezolizumab plus bevacizumab vs. sorafenib for unresectable hepatocellular carcinoma. J Hepatol. 2022 Apr;76(4):862-873. doi: 10.1016/j.jhep.2021.11.030. Epub 2021 Dec 11. PMID 34902530
- [Background] Qin S, Chen M, Cheng AL, Kaseb AO, Kudo M, Lee HC, Yopp AC, Zhou J, Wang L, Wen X, Heo J, Tak WY, Nakamura S, Numata K, Uguen T, Hsiehchen D, Cha E, Hack SP, Lian Q, Ma N, Spahn JH, Wang Y, Wu C, Chow PKH; IMbrave050 investigators. Atezolizumab plus bevacizumab versus active surveillance in patients with resected or ablated high-risk hepatocellular carcinoma (IMbrave050): a randomised, open-label, multicentre, phase 3 trial. Lancet. 2023 Nov 18;402(10415):1835-1847. doi: 10.1016/S0140-6736(23)01796-8. Epub 2023 Oct 20. PMID 37871608
- [Background] Vogel A, Meyer T, Saborowski A. IMbrave050: the first step towards adjuvant therapy in hepatocellular carcinoma. Lancet. 2023 Nov 18;402(10415):1806-1807. doi: 10.1016/S0140-6736(23)01962-1. Epub 2023 Oct 23. No abstract available. PMID 37883983
- [Background] Meyers BM, Knox JJ, Liu DM, McLeod D, Ramjeesingh R, Tam VC, Lim HJ. The evolution of immune checkpoint inhibitor combinations in advanced hepatocellular carcinoma - A systematic review. Cancer Treat Rev. 2023 Jul;118:102584. doi: 10.1016/j.ctrv.2023.102584. Epub 2023 May 27. PMID 37336142
- [Background] Leowattana W, Leowattana T, Leowattana P. Systemic treatment for unresectable hepatocellular carcinoma. World J Gastroenterol. 2023 Mar 14;29(10):1551-1568. doi: 10.3748/wjg.v29.i10.1551. PMID 36970588
- [Background] Cholankeril G, Patel R, Khurana S, Satapathy SK. Hepatocellular carcinoma in non-alcoholic steatohepatitis: Current knowledge and implications for management. World J Hepatol. 2017 Apr 18;9(11):533-543. doi: 10.4254/wjh.v9.i11.533. PMID 28469809
- [Background] Bosch FX, Ribes J, Diaz M, Cleries R. Primary liver cancer: worldwide incidence and trends. Gastroenterology. 2004 Nov;127(5 Suppl 1):S5-S16. doi: 10.1053/j.gastro.2004.09.011. PMID 15508102
- [Background] Capocaccia R, Sant M, Berrino F, Simonetti A, Santi V, Trevisani F; EUROCARE Working Group. Hepatocellular carcinoma: trends of incidence and survival in Europe and the United States at the end of the 20th century. Am J Gastroenterol. 2007 Aug;102(8):1661-70; quiz 1660, 1671. doi: 10.1111/j.1572-0241.2007.01337.x. Epub 2007 Jun 6. PMID 17555459
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines on the management of hepatocellular carcinoma. J Hepatol. 2025 Feb;82(2):315-374. doi: 10.1016/j.jhep.2024.08.028. Epub 2024 Dec 17. PMID 39690085
- [Background] Forner A, Llovet JM, Bruix J. Hepatocellular carcinoma. Lancet. 2012 Mar 31;379(9822):1245-55. doi: 10.1016/S0140-6736(11)61347-0. Epub 2012 Feb 20. PMID 22353262